CLINICAL TRIAL: NCT05597436
Title: An Expanded Access Protocol of Intravenous Trehalose Injection 90.5 mg/mL Treatment of Patients With Amyotrophic Lateral Sclerosis
Brief Title: Intermediate-Sized Expanded Access Study
Status: No longer available | Type: Expanded Access
Sponsor: Seelos Therapeutics, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: SLS-005-EAP; UF1NS131791 (NIH)
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Lou Gehrig's Disease; Trehalose; Seelos Therapeutics; SLS-005
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Trehalose

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Trehalose — Once weekly 0.75g/kg administration
  Other Names: SLS-005 Intravenous Trehalose Injection 90.5 mg/mL

SUMMARY:
This expanded access protocol is to provide access to the investigational product, SLS-005, to participants with ALS who are not eligible to participate in clinical trials.

DETAILED DESCRIPTION:
Approximately 70 participants receive a weekly infusion of SLS-005 for up to 24 weeks. There are 25 infusions over 24 weeks (first infusion occurs at the Screening/Baseline Visit). In addition to infusion visits, participants will have three scheduled in-clinic visits at Screening/Baseline, Week 3, and Week 24, and 2 phone call or telemedicine visits at Week 12 and approximately 28 days following the last dose of the investigational medical product.

ELIGIBILITY:
Inclusion Criteria:

1. Sporadic or familial ALS.
2. Age 18 years or older.
3. Cohort 1: Patients who do not qualify for any reasonably accessible ongoing clinical trial.
4. Cohort 2: Patients who have completed the open label extension (OLE) period of Regimen E of the HEALEY ALS Platform Trial and are not eligible for enrollment in another treatment regimen of the platform study.
5. Capable of providing informed consent and complying with study procedures, in the Site Investigator's (SI's) opinion.
6. Participants have established care with a physician at the specialized ALS center involved in the study and will maintain this clinical care throughout the duration of the EAP.
7. Participants must have a life expectancy of at least 6 months in SI's opinion.

Exclusion Criteria:

1. Current diagnosis or healthcare professional-recommended treatment (medication, exercise or diet) of diabetes mellitus.
2. Screening glucose >=140 mg/dl.
3. Known hypersensitivity to trehalose.
4. Current use of oral trehalose.
5. Inability for participant to return to site for weekly drug administration, until approved for home infusions.
6. Screening body weight >144 kilograms.
7. Participant with a history of any clinically significant or unstable medical condition or lab abnormality based on the SI's judgment that may interfere with assessment of the study objectives, with safety or full participation.
8. Females who are pregnant or nursing or who plan to get pregnant during the course of the EAP.
9. Females of child-bearing potential, or males, who are unwilling or unable to use highly effective methods of birth control.
10. Use of investigational treatments for ALS (as part of participation in a clinical trial or another EAP) within 5 half-lives (if known) or 30 days (whichever is longer) prior to the Screening Visit.
11. Permanent assisted ventilation (PAV), defined as more than 22 hours per day of noninvasive or invasive mechanical ventilation for more than seven consecutive days. The date of onset of PAV is the first day of the seven days.
12. Active cancer or history of cancer, except for the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin, cervical carcinoma in situ, prostatic carcinoma in situ, or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
13. Presence of unstable psychiatric disease, cognitive impairment, dementia, or substance abuse that would impair ability of the participant to provide informed consent, in the SI's opinion.
14. Patients who chose to take experimental medications and/or supplements, and that is the only reason they are not eligible for trials, won't be eligible for the EAP.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Suma Babu, MD,MPH,MBBS, Principal Investigator — Massachusetts General Hospital; James D Berry, MD,MPH, Principal Investigator — Massachusetts General Hospital; Sabrina Paganoni, MD,PhD, Principal Investigator — Massachusetts General Hospital
Locations (21):
- United States (21):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California, Irvine, Orange, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Holy Cross Hospital - Phil Smith Neuroscience Institute, Fort Lauderdale, Florida
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Sean M. Healey & AMG Center for ALS Neurological Clinical Research Institute, Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Spectrum Health/Corewell Health, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Texas Neurology, P.A.-Neal Site:769, Dallas, Texas
  - Virginia Commonwealth University Clinical Research Unit, Richmond, Virginia

REFERENCES:
- [Result] Krivickas B, Scirocco E, Giacomelli E, Sharma S, Benson M, Keegan M, Kulesa-Kelley J, Chibnik LB, Casagrande G, Heyd L, Chase M, Drake K, Mohapatra S, Hagar JL, Hasenoehrl MG, Dagostino D, Sherman AV, Leite A, Yu H, Rosenthal J, Miller T, McCaffrey A, Gwathmey K, Locatelli E, Bayat E, Heitzman D, Young E, Goyal NA, Whitesell J, Felice K, Ilieva H, Swenson A, Walk D, Alameda G, Foster L, McIlduff CE, Walsh A, Zilliox L, Ajroud-Driss S, Bodkin C, Katz J, Ladha S, Rivner M, Rosow L, Twydell P, Wasiewski W, Babu S, Berry JD, Paganoni S. Multicenter Expanded Access Protocol for Research Through Access to Trehalose in People With Amyotrophic Lateral Sclerosis. Muscle Nerve. 2025 Nov;72(5):1108-1116. doi: 10.1002/mus.70011. Epub 2025 Aug 26. PMID 40857020

DOCUMENTS (2):
  • Study Protocol (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT05597436/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT05597436/SAP_001.pdf